CLINICAL TRIAL: NCT01115777
Title: Prospective Assessment of Quality of Life (QOL) in Pediatric Patients Treated With Radiation Therapy for Brain Tumors and Non-CNS Malignancies
Brief Title: Prospective Assessment of Quality of Life (QOL) in Pediatric Patients Treated With Radiation Therapy for Brain Tumors and Non-central Nervous System (Non-CNS) Malignancies
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Torunn Yock, MD, Director, Pediatric Radiation Oncology, Massachusetts General Hospital
Other Study IDs: 2005P001629
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Brain Tumors; Non-CNS Malignancies
Keywords: Pediatric patients; treated with; radiation therapy; for brain tumors; and non-CNS malignancies
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pediatric patients treated with radiotherapy
  Interventions: Other: Quality of Life surveys completed at specified timepoints

INTERVENTIONS:
Other: Quality of Life surveys completed at specified timepoints — Quality of Life surveys (no treatment)

SUMMARY:
In recent years, remarkable advances in medical oncology, surgery, and radiology have allowed for increasing cure rates for childhood malignancies. This success has led to an emerging understanding of the kinds of effects that treatments can have on the pediatric population and how such effects can influence pediatric cancer survivor's functioning and quality of life. It has become tremendously important to assess the long-term complications due to therapy in this growing sector of survivors and to tailor our treatments so as to minimize these late effects.

The Investigators at MGH are committed to improving the delivery of radiotherapy to our patients and improving the outcome for these patients. MGH has an on-site cyclotron for proton radiotherapy in order to provide the most advanced care for patients in need. Proton therapy possesses a clinical advantage over standard photon therapy in that its optimal dose distribution delivers the bulk of radiation to the tumor site. This method spares the greatest volume of normal tissue, resulting in decreased short-term and long-term morbidity.

Through open pediatric protocols for patients treated with proton radiotherapy, the investigators aim to define and report the acute and late effects associated with treatment.

The investigators also treat a number of patients off-protocol with both proton and photon radiotherapy, and are interested in reporting these patients' QOL outcomes in conjunction with other clinical data that may be pertinent to the site of tumor treatment. This research is significant in that it will allow us to delineate the positive and negative effects of radiation treatment on patients' QOL, highlighting points of success and exposing areas that are in need of improvement. Such knowledge will be used to improve the experience of pediatric cancer survivors in the future.

The aims of this study are: 1) to prospectively collect and report the QOL outcomes in patients treated with radiotherapy and 2) to correlate the QOL data with pertinent clinical information.

DETAILED DESCRIPTION:
You will be asked to complete a series of questionnaires during your treatment and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Any patient being treated with radiation therapy with curative intent
* Patients between the ages of 2 and 25
* Patients who speak either English or Spanish
* Patients who agree to fill out the questionnaire

Exclusion Criteria:

* Patients younger than 2 years of age or over 25
* Patients receiving treatment with palliative intent
* Patients who do not wish to participate

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients coming to MGH for radiation therapy with curative intent.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2005-09; Primary Completion 2025-06 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of Quality of Life | 10 years
  Longitudinal description of quality of life outcomes in patients treated with radiation therapy

SECONDARY OUTCOMES:
Correlation of QOL data with clinical information | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Torunn Yock, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States